CLINICAL TRIAL: NCT02348541
Title: A Post-Market Clinical Follow-up Study to Investigate the Usability of the CollaGUARD Adhesion Barrier Following Hysteroscopic Adhesiolysis
Brief Title: Usability of the CollaGUARD Adhesion Barrier Following Hysteroscopic Adhesiolysis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Innocoll (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INN-CG-001
Record Dates: First submitted 2015-01-19; First posted 2015-01-28 (Estimated); Last update posted 2021-09-10 (Actual); Status verified 2021-09

CONDITIONS: Hysteroscopic Adhesiolysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CollaGUARD (Other)
  Interventions: Device: CollaGUARD

INTERVENTIONS:
Device: CollaGUARD

SUMMARY:
Assess the feasibility of CollaGUARD following Hysteroscopic Adhesiolysis.

DETAILED DESCRIPTION:
Intrauterine adhesions following gynaecological surgery is a major complication which may cause a range of severe clinical symptoms in women. IUA's can result in menstrual abnormalities, dysmenorrhea and infertility. In pregnancy, adhesions are related to miscarriage, ectopic pregnancy, abnormal placentation, premature labor and delivery and possibly birth defects.

CollaGUARD adhesion barrier is a transparent bioresorbable film approved in Europe for the prevention of postoperative adhesions in patients undergoing abdomino-pelvic laparotomy or laparoscopy.

This study will assess the feasibility of using CollaGUARD adhesion device in hysteroscopic surgery.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with intrauterine adhesions and found eligible for hysteroscopic adhesiolysis
* Willing to use additional contraception throughout study

Exclusion Criteria:

* Be pregnant or having a suspected molar pregnancy, lactating, or planning to become pregnant at any time during the study
* Has suffered or currently suffers from a gynaecological malignancy
* Has undergone a previous hysteroscopic surgery (such as removal of fibroids)

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2014-12; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Feasibility of using CollaGUARD in hysteroscopic adhesiolysis: Surgeon completed questionnaire | following initial hysteroscopy
  surgeon completed questionnaire

SECONDARY OUTCOMES:
Number of de novo adhesion and adhesion reformation | 9 weeks post initial hysteroscopy
  assessed during follow-up hysteroscopy
Change in severity of adhesions | 9 weeks post initial hysteroscopy
  European Society Gynecological Endoscopy (ESGE) classification of IUA's; modified American Fertility Society (mAFS)
Degradation of CollaGUARD | 2 weeks post initial hysteroscopy
  assessed via ultrasound

CONTACTS AND LOCATIONS:
Overall Officials: David Prior, PhD, Study Director — Sponsor GmbH
Locations (2):
- Netherlands (2):
  - Sint Lucas Andreas Ziekenhuis, Amsterdam
  - Spaarne Ziekenhuis, Hoofddorp